CLINICAL TRIAL: NCT04226118
Title: Efficacy of an Infrared Visualization Technique for the Identification of the Peripheral Venous Access Site in Patients With Cystic Fibrosis Aged 12 Years and Older
Acronym: MUCOVEINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL19_0036
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients who have a peripheral venous access by a classic procedure, without using a Vein Illumination System.
- Experimental Group (Experimental): Patients who have a peripheral venous access by a procedure using a Vein Illumination System.
  Interventions: Device: Vein Illumintion System device

INTERVENTIONS:
Device: Vein Illumintion System device — Spotting veins of a patient by use of a Vein Illumintion System device
  Arms: Experimental Group

SUMMARY:
Cystic fibrosis is a rare chronic genetic disease that mainly affects the respiratory tract and the digestive system. Their management includes multi-year intravenous antibiotic treatments and repeated venous sampling. The venous access is a source of difficulties that nurses who take care of these patients face on a daily basis. In addition, multiple attempts at punctures can induce anxiety and pain in patients. It is therefore important to limit failures.

Vein visualization technologies exist: guidance echo, portable trans lumination or infrared visualization can guide venipuncture and limit failures.

Compared with the guided echo or the portable trans lumination, the infrared visualization is easy to use and does not pose a risk for the patient. Nevertheless, studies evaluating this technique are few in chronic diseases and mainly conducted in young children.

This study aims to show that the use of a vein illumination system (VIS) should improve the peripheral venous access at the first attempt (thus limiting venous lesions) in adolescent and adult patients with cystic fibrosis, and improve comfort of the patient (pain, apprehension of the gesture).

DETAILED DESCRIPTION:
Background :

Cystic fibrosis is a rare chronic genetic disease that mainly affects the respiratory tract and the digestive system. Their management includes multi-year intravenous antibiotic treatments and repeated venous sampling. The venous access is a source of difficulties that nurses who take care of these patients face on a daily basis. In addition, multiple attempts at punctures can induce anxiety and pain in patients. It is therefore important to limit failures.

Vein visualization technologies exist: guidance echo, portable trans lumination or infrared visualization can guide venipuncture and limit failures.

Compared with the guided echo or the portable trans lumination, the infrared visualization is easy to use and does not pose a risk for the patient. Nevertheless, studies evaluating this technique are few in chronic diseases and mainly conducted in young children.

This study aims to show that the use of a vein illumination system (VIS) should improve the peripheral venous access at the first attempt (thus limiting venous lesions) in adolescent and adult patients with cystic fibrosis, and improve comfort of the patient (pain, apprehension of the gesture).

Objectives of the study :

The main objective of the study is to demonstrate that the use of a vein illumination system (VIS) for the placement of a peripheral venous line or venous sampling on the hand, forearm or fold of the elbow improves peripheral venous access (PVA) successful on the first attempt.

The secondary objectives are :

* To study the efficacy of VIS for peripheral venous access (placement of a peripheral venous line or peripheral venous sampling in the hand, forearm or elbow) on the number of attempts.
* To study the impact of the use of SIV on the patient's pain felt during the peripheral venous access procedure.
* To study the impact of VIS on patient anxiety prior to peripheral venous access.
* To describe the nurses and nursing students satisfaction with the use of the VIS device for peripheral venous access.
* To study the determinants of the success of peripheral venous access at the first attempt among the characteristics of nurses and nursing students (age, year of obtaining their diploma, experience within the cystic fibrosis ressource and competence center).
* To describe the nurses and nursing students satisfaction with the use of A-DIVA scale.

Study design The study will last 36 months. It is an open and randomized multicenter cluster study, with sequential allocation of the device (stepped wedge allocation), comparing a group of patients benefiting from a technique of locating the puncture site by a venous illumination system for a peripheral venoux access (hand, forearm, fold of the elbow) to a group of patients whose veins are identified according to the usual modality of a peripheral venoux access. The cluster is defined by the Cystic Fibrosis Resource and Competence Center (CRCM).

Expected results

For the patients, the use of a venous illumination system device during the peripheral venous access should facilitate the success of the gesture on the first attempt, allowing to :

* Reduce their pain due to multiple attempts.
* Reduce their anxiety associated with peripheral venous access.
* Preserve their venous capital This could have an impact on their care, such as making it easier to consult for them and being less anxious about peripheral venous access.

For the nurses, using a venous illimunation system device could

* Reduce their apprehension of peripheral venous access gesture
* Save their time with fewer peripheral venous access are repeated. It is considered that this technique will be distributed to all Cytic Fibrosis Ressource and Competence Centers (CRCM) in order to improving the comfort of the chronically ill patient with repeated blood tests and intravenous treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cystic fibrosis aged 12 years and over
* Cystic Fibrosis diagnosis has been confirmed by a positive sweat test and/or 1 to 2 genetic mutations
* Patients requiring peripheral venous access (hand, forearm, or more of the elbow) for intravenous infusion with epicranial or short catheter, or for a blood sample
* Patients who have a score of 4 or higher on the A-DIVA scale (self-administered questionnaire completed by the IDE assessing the difficulty of peripheral venous access on a Likert scale from 0 to 8)
* Patients informed in writing of the terms of the study and provided written informed consent to participate (consent of the person in charge of parental authority if the patient is a minor).
* Patients affiliated to a social security system

Exclusion Criteria:

* Patient who has already participated in the study
* Patients who have a central venous approach
* Patients who have a venous approach of the midline type
* Patients taken care of for vital emergency
* Patient deprived of liberty or placed under tutorship or curatorship

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients for whom peripheral venous access was performed from the first attempt. | at time of peripheral venous access

SECONDARY OUTCOMES:
Number of attempts to place a peripheral venous line or perform peripheral venous | at time of peripheral venous access
Average pain score on Visual Analogue Scale (VAS) after successful peripheral venous access act. | at most 10 min after the venous act
Average anxiety score on State-Trait Anxiety Inventory (STAI-Y) | at most 10 min before the venous act
Proportion of nurses and nursing student satisfied by the use of a vein illumination system | at the end of the study ( at 14 months)

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CRCM mixte de Giens, Giens
  - Hôpital Nord - CRCM adulte Marseille, Marseille
  - Hôpital enfant la Timone - CRCM pédiatrique Marseille, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpital Pasteur - CRCM adulte Nice, Nice
  - Hôpital Lenval - CRCM pédiatrique Nice, Nice